CLINICAL TRIAL: NCT02591901
Title: Prevention of Recurrent Symptomatic Urinary Tract Infections in Participants With Chronic Neurogenic Bladder Dysfunction: A Mixed Method Study
Brief Title: Preventing UTIs in Chronic Neurogenic Bladder Dysfunction (Mix Methods)
Acronym: PReSuTINeB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Oxford Clinical Trials Research Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RXQ/648
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: UTI; Neurogenic Bladder; Antibiotic Resistance
Keywords: Spinal Cord Injuries; Multiple Sclerosis; Transverse Myelitis; Neurogenic Bladder Dysfunction; Feasibility Study; Urinary Tract Infection
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries; Multiple Sclerosis; Myelitis, Transverse; Urinary Tract Infections | interventions — OM 89

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uro Vaxom (Experimental): Uro Vaxom, Once daily for 3 months
  Interventions: Drug: Uro vaxom
- Placebo (Placebo Comparator): Placebo identical to main drug in shape and form
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: Uro vaxom — Prevention of recurrent symptomatic lower urinary tract infections
  Other Names: OM-89
  Arms: Uro Vaxom
Other: Placebo comparator — Placebo comparator
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Due to the damage caused to the spinal cord, patients with spinal cord injury, cauda equina syndrome, multiple sclerosis and transverse myelitis may encounter loss of bladder function, which in turn can lead to a debilitating and costly complication: Urinary Tract Infections (UTIs). Given that these patients with loss of bladder function do not normally feel symptoms like pain - as would be the case in otherwise healthy persons - there is no clear agreement among experts on which signs and symptoms are indicative of a UTI. Although strong evidence is lacking, antibiotics have been widely used for prevention of recurrent UTIs in patients with loss of bladder function. However, this approach is now being questioned as antibiotic resistance has become a world-wide health concern. Policy makers recently stressed the importance of research into alternative preventative treatments. The use of immunotherapy is one such an alternative approach, which works by stimulating the body's immune system. One of these immunotherapy is a Uro-Vaxom® oral capsule which consists of inactivated traces of the bacteria that normally cause at least 83% of UTIs in patients with loss of bladder function. Previous studies show that Uro-Vaxom® resulted in a significant reduction of UTIs in otherwise healthy patients, as well as being safe to use. Before investigating the effects of this promising new immunotherapy, this proposed study aims to clarify two crucial issues. First, after reviewing the literature and appraising patients', carers' and healthcare professionals' experiences, the aim is to reach an agreement on how to measure a symptomatic UTI in patients with loss of bladder function that results from a spinal cord lesion. Second, using Uro-Vaxom® Investigators aim to conduct a smallscale, placebo-controlled trial with 48 participants to investigate the feasibility of carrying out a larger trial on prevention of symptomatic UTI in such patients.

DETAILED DESCRIPTION:
Each year in the UK 1,200 people sustain a spinal cord injury, 600 people will be diagnosed with cauda equina syndrome, 6,000 with multiple sclerosis and 300 with transverse myelitis. These four patient groups all suffer from neurological disorders of the spinal cord, resulting in loss of normal bladder function known as neurogenic bladder dysfunction. This in turn can lead to urinary tract infections (UTIs). UTIs are a commonly recurring and debilitating complication, with spinal patients experiencing 2.5 episodes per patient per year on average. This not only results in 16% of hospital readmissions and costs of care of up to £125 million spent by the NHS on treating UTIs every year, but also has a dramatic impact on patients' quality of life.

A recent NICE guideline highlighted the methodological difficulties of research into the prevention of UTIs in patients with neurogenic bladder dysfunction. Given that this group of patients normally do not feel symptoms like 'pain' and 'a frequent urge to urinate', it can be difficult to distinguish between bladder colonisation (asymptomatic bacteriuria) and true infection (a symptomatic UTI). To date, there is no clear agreement among experts on which signs and symptoms are indicative of a symptomatic UTI. Although strong evidence is lacking, antibiotics have been widely used for the prevention of recurrent UTIs in patients with neurogenic bladder dysfunction. However, this approach is now being called into question as antibiotic resistance has become a world-wide health concern.

In the recently published 'UK Five Year Antimicrobial Resistance Strategy', policy makers stressed the importance of research into alternative preventative treatments. Immunotherapy potentially offers such a (cost-) effective alternative to antibiotic therapy for UTI management. At least 83% of community-acquired complicated UTIs are caused by Escherichia coli (E. coli). Uro-Vaxom® (OM-Pharma, Switzerland) is an orally administered, bacterial vaccine which consists of a 6mg lyophilised (heat-inactivated) mix of E. coli membrane glycoproteins.

Previous studies showed that Uro-Vaxom® resulted in a significant reduction of UTIs in otherwise healthy women with recurrent cystitis, as well as being safe to use.

Before investigating the effects of this promising new vaccine in patients with neurogenic bladder dysfunction, two crucial issues will need to be clarified. First, consensus must be reached on how to measure a symptomatic UTI in this group of patients. Second, the feasibility of carrying out a larger, definitive randomised controlled trial on the prevention of symptomatic UTI in patients with neurogenic bladder dysfunction must be established. The central aim of the proposed mixed method study is to clarify these two key methodological and feasibility issues.

In the first stage of this study is to carry out qualitative interviews to explore patient experiences and views of symptoms and signs associated with a UTI. These results, combined with findings from a literature review, will enable the design of a quantitative patient survey which will be distributed by four service user organisations to people with neurogenic bladder dysfunction. Finally, taking the results from all preceding stages, a final definition, or algorithm, will be discussed before and during a consensus meeting.

In the second stage of this study, a small-scale parallel, double-blinded, randomised, placebo-controlled, multicentre trial will be conducted to investigate the feasibility of carrying out a larger well-powered study on the prevention of symptomatic UTI in patients with neurogenic bladder dysfunction. Forty-eight patients will be randomly assigned treatment with Uro-Vaxom®, or placebo, for 3 months and followed-up for a further 3 months.

This is to expose any pitfalls or areas requiring re-designing, such as logistics, recruitment and compliance rates, in order to refine the protocol of a definitive clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of spinal cord injury, multiple sclerosis, transverse myelitis or cauda equina damage;
* Have had the diagnosis of the spinal pathology for at least 12 months;
* Have not had any significant changes in the underlying condition for 12 weeks
* Be living in the community (not in residential care)
* Aged 18 to 75 years
* Have had at least three urinary tract infection episodes treated using anti-biotics over the preceding 12 months;
* If a woman of child-bearing age, is willing to use contraception for the duration of the study
* Having the mental capacity to give informed consent

Exclusion Criteria:

* Have had surgical alterations to the bladder, excluding supra-pubic catherisation.
* Known hypersensitivity to the active principle or to any of the excipients of Uro-Vaxom®
* Being unwilling to take a product containing gelatin (e.g. vegetarians)

  * recruitment can be postponed until antibiotics have not been used for a period of 14 days and symptoms of a UTI have subsided

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-09-21 (Actual)

PRIMARY OUTCOMES:
Checklist or consensus guideline which can be used to measure a symptomatic urinary tract infection and Practicality of carrying out a definitive randomised controlled clinical study | 23 months

SECONDARY OUTCOMES:
Number of participants willing to participate | 14 months
Number of successfully collected urine samples via courier | 14 months
Drug compliance | 14 months
  Measured by the number of un-used drug packs that the participants will return upon each hospital visit

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Belci, DMS MSc MRCS FRCP, Principal Investigator — Stoke Mandeville Hospital
Locations (2):
- United Kingdom (2):
  - Stoke Mandeville Hospital, Aylesbury, Buckinghamshire
  - Oxford Centre for Enablement, Oxford, Oxfordshire

REFERENCES:
- [Background] Esclarin De Ruz A, Garcia Leoni E, Herruzo Cabrera R. Epidemiology and risk factors for urinary tract infection in patients with spinal cord injury. J Urol. 2000 Oct;164(4):1285-9. PMID 10992382
- [Background] D'Hondt F, Everaert K. Urinary tract infections in patients with spinal cord injuries. Curr Infect Dis Rep. 2011 Dec;13(6):544-51. doi: 10.1007/s11908-011-0208-6. PMID 21853416
- [Background] Manack A, Motsko SP, Haag-Molkenteller C, Dmochowski RR, Goehring EL Jr, Nguyen-Khoa BA, Jones JK. Epidemiology and healthcare utilization of neurogenic bladder patients in a US claims database. Neurourol Urodyn. 2011 Mar;30(3):395-401. doi: 10.1002/nau.21003. Epub 2010 Sep 29. PMID 20882676
- [Background] Street JT, Noonan VK, Cheung A, Fisher CG, Dvorak MF. Incidence of acute care adverse events and long-term health-related quality of life in patients with TSCI. Spine J. 2015 May 1;15(5):923-32. doi: 10.1016/j.spinee.2013.06.051. Epub 2013 Aug 24. PMID 23981816
- [Background] Morawietz C, Moffat F. Effects of locomotor training after incomplete spinal cord injury: a systematic review. Arch Phys Med Rehabil. 2013 Nov;94(11):2297-308. doi: 10.1016/j.apmr.2013.06.023. Epub 2013 Jul 9. PMID 23850614
- [Background] Lavy C, James A, Wilson-MacDonald J, Fairbank J. Cauda equina syndrome. BMJ. 2009 Mar 31;338:b936. doi: 10.1136/bmj.b936. No abstract available. PMID 19336488
- [Background] Gupta A, Taly AB, Srivastava A, Murali T. Non-traumatic spinal cord lesions: epidemiology, complications, neurological and functional outcome of rehabilitation. Spinal Cord. 2009 Apr;47(4):307-11. doi: 10.1038/sc.2008.123. Epub 2008 Oct 21. PMID 18936767
- [Background] West TW. Transverse myelitis--a review of the presentation, diagnosis, and initial management. Discov Med. 2013 Oct;16(88):167-77. PMID 24099672
- [Background] Rubin SM. Management of multiple sclerosis: an overview. Dis Mon. 2013 Jul;59(7):253-60. doi: 10.1016/j.disamonth.2013.03.012. No abstract available. PMID 23786659
- [Background] Ersoz M, Tunc H, Akyuz M, Ozel S. Bladder storage and emptying disorder frequencies in hemorrhagic and ischemic stroke patients with bladder dysfunction. Cerebrovasc Dis. 2005;20(5):395-9. doi: 10.1159/000088670. Epub 2005 Oct 3. PMID 16205058
- [Background] Benevento BT, Sipski ML. Neurogenic bladder, neurogenic bowel, and sexual dysfunction in people with spinal cord injury. Phys Ther. 2002 Jun;82(6):601-12. PMID 12036401
- [Background] Jamison J, Maguire S, McCann J. Catheter policies for management of long term voiding problems in adults with neurogenic bladder disorders. Cochrane Database Syst Rev. 2013 Nov 18;2013(11):CD004375. doi: 10.1002/14651858.CD004375.pub4. PMID 24249436
- [Background] Sedor J, Mulholland SG. Hospital-acquired urinary tract infections associated with the indwelling catheter. Urol Clin North Am. 1999 Nov;26(4):821-8. doi: 10.1016/s0094-0143(05)70222-6. PMID 10584622
- [Background] Khatri B, Basnyat S, Karki A, Poudel A, Shrestha B. Etiology and antimicrobial susceptibility pattern of bacterial pathogens from urinary tract infection. Nepal Med Coll J. 2012 Jun;14(2):129-32. PMID 23671963
- [Background] Cai T, Mazzoli S, Mondaini N, Meacci F, Nesi G, D'Elia C, Malossini G, Boddi V, Bartoletti R. The role of asymptomatic bacteriuria in young women with recurrent urinary tract infections: to treat or not to treat? Clin Infect Dis. 2012 Sep;55(6):771-7. doi: 10.1093/cid/cis534. Epub 2012 Jun 7. PMID 22677710
- [Background] Willing BP, Russell SL, Finlay BB. Shifting the balance: antibiotic effects on host-microbiota mutualism. Nat Rev Microbiol. 2011 Apr;9(4):233-43. doi: 10.1038/nrmicro2536. Epub 2011 Feb 28. PMID 21358670
- [Background] Werndle MC, Zoumprouli A, Sedgwick P, Papadopoulos MC. Variability in the treatment of acute spinal cord injury in the United Kingdom: results of a national survey. J Neurotrauma. 2012 Mar 20;29(5):880-8. doi: 10.1089/neu.2011.2038. Epub 2011 Oct 26. PMID 21939394
- [Background] Plowman, R., Graves, N., Griffin, M., Swan, A., Cookson, B., Taylor, L. 1999. The socio-economic burden of healthcare associated infection. PHLS.
- [Background] National Clinical Guideline Centre (UK). Urinary Incontinence in Neurological Disease: Management of Lower Urinary Tract Dysfunction in Neurological Disease. London: Royal College of Physicians (UK); 2012 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK132831/ PMID 23638496
- [Background] Karlowsky JA, Hoban DJ, Decorby MR, Laing NM, Zhanel GG. Fluoroquinolone-resistant urinary isolates of Escherichia coli from outpatients are frequently multidrug resistant: results from the North American Urinary Tract Infection Collaborative Alliance-Quinolone Resistance study. Antimicrob Agents Chemother. 2006 Jun;50(6):2251-4. doi: 10.1128/AAC.00123-06. PMID 16723598
- [Background] Schito GC, Naber KG, Botto H, Palou J, Mazzei T, Gualco L, Marchese A. The ARESC study: an international survey on the antimicrobial resistance of pathogens involved in uncomplicated urinary tract infections. Int J Antimicrob Agents. 2009 Nov;34(5):407-13. doi: 10.1016/j.ijantimicag.2009.04.012. Epub 2009 Jun 7. PMID 19505803
- [Background] Manges AR, Johnson JR, Foxman B, O'Bryan TT, Fullerton KE, Riley LW. Widespread distribution of urinary tract infections caused by a multidrug-resistant Escherichia coli clonal group. N Engl J Med. 2001 Oct 4;345(14):1007-13. doi: 10.1056/NEJMoa011265. PMID 11586952
- [Background] Brumbaugh AR, Mobley HL. Preventing urinary tract infection: progress toward an effective Escherichia coli vaccine. Expert Rev Vaccines. 2012 Jun;11(6):663-76. doi: 10.1586/erv.12.36. PMID 22873125
- [Background] Naber KG, Cho YH, Matsumoto T, Schaeffer AJ. Immunoactive prophylaxis of recurrent urinary tract infections: a meta-analysis. Int J Antimicrob Agents. 2009 Feb;33(2):111-9. doi: 10.1016/j.ijantimicag.2008.08.011. Epub 2008 Oct 28. PMID 18963856
- [Background] Schmidhammer S, Ramoner R, Holtl L, Bartsch G, Thurnher M, Zelle-Rieser C. An Escherichia coli-based oral vaccine against urinary tract infections potently activates human dendritic cells. Urology. 2002 Sep;60(3):521-6. doi: 10.1016/s0090-4295(02)01767-3. PMID 12350510
- [Background] Bauer HW, Alloussi S, Egger G, Blumlein HM, Cozma G, Schulman CC; Multicenter UTI Study Group. A long-term, multicenter, double-blind study of an Escherichia coli extract (OM-89) in female patients with recurrent urinary tract infections. Eur Urol. 2005 Apr;47(4):542-8; discussion 548. doi: 10.1016/j.eururo.2004.12.009. Epub 2005 Jan 21. PMID 15774256
- [Background] Magasi P, Panovics J, Illes A, Nagy M. Uro-Vaxom and the management of recurrent urinary tract infection in adults: a randomized multicenter double-blind trial. Eur Urol. 1994;26(2):137-40. doi: 10.1159/000475363. PMID 7957468
- [Background] Schulman CC, Corbusier A, Michiels H, Taenzer HJ. Oral immunotherapy of recurrent urinary tract infections: a double-blind placebo-controlled multicenter study. J Urol. 1993 Sep;150(3):917-21. doi: 10.1016/s0022-5347(17)35648-3. PMID 8345609
- [Background] Tammen H. Immunobiotherapy with Uro-Vaxom in recurrent urinary tract infection. The German Urinary Tract Infection Study Group. Br J Urol. 1990 Jan;65(1):6-9. doi: 10.1111/j.1464-410x.1990.tb14649.x. PMID 2178724
- [Background] Richie, J. and Spencer, L. Qualitative data analysis for applied policy research. In Analysing Qualitative Data. (eds A.Bryman and R.Burgess). 1994:173-194. London: Routledge
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Cardenas DD, Ditunno J, Graziani V, Jackson AB, Lammertse D, Potter P, Sipski M, Cohen R, Blight AR. Phase 2 trial of sustained-release fampridine in chronic spinal cord injury. Spinal Cord. 2007 Feb;45(2):158-68. doi: 10.1038/sj.sc.3101947. Epub 2006 Jun 13. PMID 16773037